CLINICAL TRIAL: NCT04193046
Title: A Prospective, Multicenter Study for the Identification of Biomarker Signatures for the Early Detection of Pulmonary Hypertension (PH)
Brief Title: A Study for the Identification of Biomarker Signatures for Early Detection of Pulmonary Hypertension (PH)
Acronym: CIPHER
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR108723; NAPUH0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with PH and non-PH (Other): Blood samples will be collected for biomarker analysis from new (incident) and existing (prevalent) participants who undergo right heart catheterization (RHC). Participants will be categorized into non-PH or PH based on the results of the RHC and those who are found to have PH will be further classified into the different groups of PH. A transthoracic echocardiography (TTE) will be performed if not done previously.
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Prevalent (existing) and incident (new) participants who are found to either have PH or not by RHC will provide blood sample for the establishment of a biomarker signature of PH.

SUMMARY:
The primary purpose of this study is to identify and develop biomarker signatures based on circulating micro ribonucleic acid (RNA) in the blood samples associated with high risk of pulmonary hypertension (PH) to assist in the diagnosis of PH; to estimate the sensitivity, specificity, positive predictive value, and negative predictive value of the biomarker signatures in identifying participants with PH by comparing the biomarker signatures to right heart catheterization (RHC) and to compare the sensitivity, specificity, positive predictive value, and negative predictive value of the biomarker signatures with the sensitivity, specificity, positive predictive value, and negative predictive value of transthoracic echocardiogram (TTE) in identifying participants with PH documented by RHC.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone an right heart catheterization (RHC) within 18 months (prevalent PH participants) or 6 months (prevalent non-PH participants) or have undergone or planned RHC within 6 weeks (incident participants). The results of the incident RHC (incident participants) or the most recent RHC (prevalent participants) will be used to classify the participant in one of the above study population categories
* Medically stable on the basis of physical examination, medical history and vital signs performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Must provide an Informed Consent Form (ICF) (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Must provide a separate informed consent (or their legally-acceptable representative must sign) if he or she agrees to provide an optional (deoxyribonucleic acid [DNA]) sample for research (where local regulations permit). Refusal to give consent for the optional (DNA) research sample does not exclude a participant from participation in the study

Exclusion Criteria:

* Participants requiring renal dialysis
* History of lung or heart transplant (waiting list status or consideration of enlisting is allowed)
* Severe left ventricular dysfunction: Left ventricular ejection function less then (<) 35 percent (%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 907 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Expression Levels of miRNAs Biomarkers | Day 1
  Blood samples will be collected for micro Ribonucleic acid (miRNA) assay by qPCR to identify a biomarker signature for the early detection of pulmonary hypertension (PH).
Biomarker signatures for miRNA | Day 1
  Blood will be collected for miRNA to identify a biomarker signature(s) for detection of participants at high risk of PH.
Biomarker Signature Performance in Identifying Participants with PH | Day 1
  Biomarker signature performance will be evaluated by estimating sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the biomarker signatures documented by RHC for identifying participants with PH.
Comparison of Performance of Biomarker Signatures and Transthoracic Echocardiogram (TTE) Based on Sensitivity, Specificity, Positive Predictive Value, and Negative Predictive Value | Day 1
  The performance of the biomarkers signatures will be compared to the performance of TTE to identify participants with PH documented by RHC via sensitivity, specificity, positive predictive value, and negative predictive value. The sensitivity/specificity of the tests will be compared using McNemar's test.

SECONDARY OUTCOMES:
Area Under ROC Curve in Participants with PH who are Receiving Therapies Versus not Receiving drug Therapy | Day 1
  Performance of the biomarker signatures will be assessed using ROC curve in participants with PH who are receiving pulmonary arterial hypertension-specific drug therapies versus participants who are not receiving any drug therapy.
Area Under ROC Curve in Participants with PAH, CTEPH, Isolated pre-Capillary and post-Capillary PH | Day 1
  Performance of the biomarker signatures will be assessed using ROC curve in participants with pulmonary arterial hypertension (PAH), chronic thromboembolic pulmonary hypertension (CTEPH), isolated pre-capillary and post-capillary PH.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (49):
- United States (16):
  - University of Southern California, Los Angeles, California
  - University Of Colorado Cardiac And Vascular Center, Aurora, Colorado
  - Ascension St. Vincent's Lung Institute, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University Of Iowa - Hospitals & Clinics, Iowa City, Iowa
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Pulmonary Health Physicians, PC, Liverpool, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - The Houston Methodist Research Institute, Houston, Texas
  - Pulmonary Associates Of Richmond, Richmond, Virginia
- Belgium (2):
  - ULB Erasme Ziekenhuis, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- France (5):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Hôpital Cardiologique - Chru Lille, Lille
  - CHU de Montpellier - Arnaud de Villeneuve, Montpellier
  - Hopital Larrey CHU de Toulouse, Toulouse
- Germany (7):
  - Universitatsklinikum Bonn, Bonn
  - Universitätsklinikum Carl Gustav Carus Medizinische Klinik und Poliklinik 1-Pneumologie, Dresden
  - Universitaetsklinikum Giessen, Giessen
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhaus
  - Universitätsklinikum Jena Klinik für Innere Medizin I, Jena
  - Universitatsklinikum Schleswig Holstein, Lübeck
- VUMC Amsterdam, Amsterdam, Netherlands
- Poland (3):
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego, Lublin
  - Europejskie Centrum Zdrowia Otwock Sp z o o, Otwock
  - Samodzielny Publiczny Szpital Kliniczny nr 2 PUM, Szczecin
- Spain (6):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen de La Salud, Toledo
- Ukraine (4):
  - CNE 'Cherkasy Regional Cardiological Center of Cherkasy Regional Council', Cherkasy
  - CE 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiosurgery', Dnipro
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - SI 'National Institute of Phtisiology and Pulmonology n.a. F.G. Yanovsky of NAMS of Ukraine', Kyiv
- United Kingdom (5):
  - Royal United Hospital, Bath
  - National Waiting Times Centre Board Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No